CLINICAL TRIAL: NCT07370506
Title: Efficacy of Telmisartan in Preventing Doxorubicin-induced Cardiotoxicity in Breast Cancer Patients
Brief Title: Telmisartan for Prevention of Doxorubicin-Induced Cardiotoxicity in Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mennatullah Galal Ahmed Barakat, Teaching Assistant (Demonstrator) of Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2467R4
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Doxorubicin Induced Cardiomyopathy
Keywords: Telmisartan; Anthracycline Cardiotoxicity; Troponin; NT-proBNP; Cardioprotection
MeSH Terms: conditions — Breast Neoplasms | interventions — Telmisartan; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telmisartan Group (Experimental): Participants receiving telmisartan in addition to standard doxorubicin-based chemotherapy.
  Interventions: Drug: Telmisartan; Drug: Doxorubicin (DOX)
- Control Group (Active Comparator): Participants receiving standard doxorubicin-based chemotherapy without telmisartan.
  Interventions: Drug: Doxorubicin (DOX)

INTERVENTIONS:
Drug: Telmisartan — Telmisartan administered orally once daily as cardioprotective therapy during doxorubicin-based chemotherapy.
  Arms: Telmisartan Group
Drug: Doxorubicin (DOX) — Standard doxorubicin-based chemotherapy according to institutional protocol.

SUMMARY:
This study aims to evaluate the efficacy and safety of telmisartan as a cardioprotective agent in patients receiving doxorubicin-based chemotherapy, with the goal of reducing treatment-associated cardiotoxicity, optimizing therapeutic outcomes, and facilitating the safer administration of anthracycline regimens.

DETAILED DESCRIPTION:
Doxorubicin remains one of the most effective chemotherapeutic agents for the treatment of a wide range of solid tumors and hematological malignancies. However, its clinical use is limited by dose-dependent cardiotoxicity, which may manifest as subclinical myocardial injury, left ventricular dysfunction, and progression to heart failure. The mechanisms underlying doxorubicin-induced cardiotoxicity are multifactorial, with oxidative stress recognized as a central pathway contributing to reactive oxygen species (ROS) generation, mitochondrial dysfunction, and cardiomyocyte injury. These effects highlight the need for strategies to reduce cardiovascular complications associated with doxorubicin therapy without compromising anticancer efficacy.

Telmisartan, an angiotensin II type 1 receptor blocker (ARB), has demonstrated pharmacological effects beyond blood pressure control. Preclinical studies suggest that telmisartan may reduce oxidative stress, improve endothelial function, and preserve mitochondrial integrity, partly through modulation of peroxisome proliferator-activated receptor gamma (PPAR-γ) pathways. These effects may contribute to attenuation of cardiac remodeling and myocardial injury. Despite these observations, clinical evidence evaluating telmisartan for the prevention of doxorubicin-induced cardiotoxicity remains limited and inconclusive. Recent in vitro findings also indicate that telmisartan may enhance doxorubicin-induced apoptosis and cytotoxic efficacy in cancer cell lines. These findings raise the possibility that telmisartan could exert both cardioprotective and chemosensitizing effects.

Considering this evidence gap, the present study is designed to investigate the cardioprotective role of telmisartan in patients undergoing doxorubicin-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer.
* Age ≥18 & ≤ 65 years.
* Newly diagnosed, chemotherapy-naïve patients.
* Baseline echocardiogram showing left ventricular ejection fraction (LVEF) ≥55%.

Exclusion Criteria:

* Presence of hypersensitivity to telmisartan.
* History of cardiovascular disease (e.g., congestive heart failure, ischemic heart disease, arrhythmia).
* Patients with any chronic liver or renal dysfunction; inflammatory diseases; autoimmune disease; acute cardiovascular events, eating disorders (anorexia, bulimia) or gastrointestinal disorders.
* Baseline blood pressure ≥ 160/100 mmHg
* Current or prior use of ARBs/ACE inhibitors
* Current participation in another clinical trial within the past 30 days.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline to end of chemotherapy (approximately 12-18 weeks)
  The primary outcome is the absolute change in left ventricular ejection fraction (LVEF) from baseline to the end of doxorubicin-based chemotherapy, assessed by echocardiography.

SECONDARY OUTCOMES:
Change in High-Sensitivity Cardiac Troponin T (hs-cTnT) Levels | Baseline (pre-chemotherapy) to end of chemotherapy (approximately 12-18 weeks)
  Measurement of serum hs-cTnT at baseline and at the end of doxorubicin-based chemotherapy to assess myocardial injury and cardiac stress in patients receiving telmisartan or standard care.
Change in N-terminal pro-B-type Natriuretic Peptide (NT-proBNP) Levels | Baseline to end of chemotherapy (approximately 12-18 weeks)
  Measurement of serum NT-proBNP at baseline and at the end of doxorubicin-based chemotherapy. Any increase from baseline indicates early ventricular strain or subclinical heart failure in patients receiving telmisartan or standard care.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seino Y, Takahashi H, Fukumoto H, Utsumi K, Hirai Y. Cardiovascular manifestations of Fabry disease and the novel therapeutic strategies. J Nippon Med Sch. 2005 Oct;72(5):254-61. doi: 10.1272/jnms.72.254. PMID 16247224
- [Background] Taniguchi N. From the gamma-glutamyl cycle to the glycan cycle: a road with many turns and pleasant surprises. J Biol Chem. 2009 Dec 11;284(50):34469-78. doi: 10.1074/jbc.X109.023150. Epub 2009 Oct 19. No abstract available. PMID 19840938
- [Background] Arciuli J, Simpson IC. Statistical learning is lasting and consistent over time. Neurosci Lett. 2012 May 31;517(2):133-5. doi: 10.1016/j.neulet.2012.04.045. Epub 2012 Apr 25. PMID 22561650
- [Background] Simeunovic B, Strbenc M, Bavdek SV. Position and histological structure of the testes in the brown hare (Lepus europaeus) during seasonal regression and recrudescence. Anat Histol Embryol. 2000 Apr;29(2):73-82. doi: 10.1046/j.1439-0264.2000.00233.x. PMID 10932383
- [Background] Banegas JR, Segura J, Ruilope LM, Luque M, Garcia-Robles R, Campo C, Rodriguez-Artalejo F, Tamargo J; CLUE Study Group Investigators. Blood pressure control and physician management of hypertension in hospital hypertension units in Spain. Hypertension. 2004 Jun;43(6):1338-44. doi: 10.1161/01.HYP.0000127424.59774.84. Epub 2004 Apr 26. PMID 15117908